CLINICAL TRIAL: NCT03906045
Title: A Phase I, Single-Dose, Gamma Scintigraphy Study to Assess the Pulmonary Deposition of Technetium-99m Radiolabelled Budesonide, Glycopyrronium and Formoterol Fumarate MDI in Patients With Moderate to Severe/Very Severe COPD.
Brief Title: A Scintigraphy Study of PT010 in COPD Patients
Acronym: RD708/34000
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5980C00020
Record Dates: First submitted 2019-03-25; First posted 2019-04-08 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; scintigraphy; budesonide; glycopyrronium; formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This will be a single-dose study to assess the pulmonary deposition of Radiolabelled BGF MDI following administration in male and female patients with moderate to severe/very severe COPD. SAEs will be recorded from the time of signing of informed consent form to Post-study Follow-up phone call. Non-serious AEs will be collected from the first dose on Day 1 to Post-study Follow-up phone call. Study drug will be administered by inhalation.
  The study will comprise of a Screening Visit, followed by a single Treatment Period and a Post-study Follow-up phone call.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): 10 patients with moderate COPD and 10 patients with severe/very severe COPD inhale BGF followed by a breath hold of up to 10 seconds.
  Interventions: Drug: BGF-MDI

INTERVENTIONS:
Drug: BGF-MDI — Budesonide, Glycopyrronium and Formoterol Fumarate.

SUMMARY:
This study is a single treatment period, single dose gamma scintigraphy study investigating the deposition in the lungs of a Budesonide, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (BGF-MDI). This study will be investigating how the drug (known as PT010) is distributed in the lungs of Chronic Obstructive Pulmonary Disease (COPD) patients (with moderate to very severe COPD) following a maximal 10 second breath hold. This inhaler is intended to be used in the treatment of COPD, which is a group of diseases which cause lung problems and difficulty breathing. PT010 is a new combination product of 3 marketed drugs called Glycopyrronium, Formoterol Fumarate and Budesonide.

DETAILED DESCRIPTION:
This will be a single-dose study to assess the pulmonary deposition of Radiolabelled BGF MDI following administration in male and female patients with moderate to severe/very severe COPD. Serious Adverse Events (SAEs) will be recorded from the time of signing of informed consent form to Post-study Follow-up phone call. Non-serious Adverse Events (AEs) will be collected from the first dose on Day 1 to Post-study Follow-up phone call. Study drug will be administered by inhalation.

The study will comprise of a Screening Visit, followed by a single Treatment Period and a Post-study Follow-up phone call. The Treatment Period will be from the afternoon before (Day 1) until 4 hours (h) post dose (Day 1). Patients will arrive at the Clinical Unit on Day 1. Patients will withhold their regular COPD medication in the morning of Day 1 and instead be given short-acting Ventolin Hydrofluoroalkane (HFA) and Atrovent HFA which may be used up to (but not within) 6 h prior to dosing. Investigational Product (IP) will be administered on the afternoon of Day 1 fasted (after a fast of at least 2 h) and patients will be discharged 4 h post dose (Day 1), provided there are no ongoing safety concerns. During the treatment period, patients will also undergo a Krypton-81m (81mKr) gas ventilation imaging scan and a Cobalt-57 (57Co) transmission scan. SAEs will be evaluated from the time of signing the informed consent form and up to the Post-study Follow-up phone call, non-serious AEs will be evaluated from Day 1 following IP dose and up to the Post-study Follow-up phone call. Approximately 20 patients (10 per cohort) will be enrolled for at least 16 to complete the study:

* Approximately 10 patients with moderate COPD (Forced Expiratory Volume in 1 Second (FEV1) ≥50-<80% of predicted normal), for at least 8 completed patients.
* Approximately 10 patients with severe/very severe COPD (FEV1 <50% of predicted normal), for at least 8 completed patients.

At the time of dosing, patients will be required to perform 2 inhalations (after priming) under the supervision of an Investigator. Immediately following each inhalation, patients will perform a maximal breath-hold, up to 10 s, prior to exhaling into an exhalation filter. Once the second breath hold and exhalation has been performed, patients will rinse their mouth with water and expel the washings for collection. Patients will then swallow bread and water.

Thereafter, posterior and anterior views of the lungs and stomach, and a lateral head and neck view will be recorded using a gamma camera. All images will be of a maximum of 200 s in duration. Images will also be acquired of the exhalation filter and collected mouth washings. Mass balance calculations will be undertaken to determine the fraction of the emitted dose delivered to the lungs of the patients. The distribution pattern of radiolabel within the lungs will be described in terms of a ratio of radioactive counts in different lung regions, after accounting for differences in regional lung volumes.

ELIGIBILITY:
Main Inclusion Criteria:

* Males and females at least 40 years of age and no older than 80 years.
* Patients with diagnosis of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) [1].

  * Post bronchodilator (BD) FEV1 / Forced Vital Capacity (FVC) ratio must be < 0.70.
  * Post BD FEV1 must be < 80% predicted.
* All patients must be receiving 1 or more inhaled maintenance therapies, including at least 1 long-acting bronchodilator, for the management of their COPD for at least 4 weeks prior to the Screening Visit.
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking. [Number of pack-years = (number of cigarettes per day/20) x number of years smoked (e.g. 20 cigarettes per day for 10 years or 10 cigarettes per day for 20 years represent 10 pack-years)].

Main Exclusion Criteria:

* Any significant disease or disorder (e.g. including but not limited to gastrointestinal, hepatic, renal/urinary tract, haematological, neurological, musculoskeletal, endocrine, metabolic, eye, psychiatric which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results of the study.
* Respiratory:

Current diagnosis of asthma, in the opinion of the Investigator. COPD due to α1-Antitrypsin Deficiency. Sleep apnoea that, in the opinion of the Investigator, is uncontrolled. Other Respiratory Disorders: known active tuberculosis, lung cancer, cystic fibrosis, significant bronchiectasis (high resolution computerised tomography [CT] evidence of bronchiectasis that causes repeated acute exacerbations), immune deficiency disorders, severe neurological disorders affecting control of the upper airway, sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or pulmonary thromboembolic disease. Note: allergic rhinitis is not exclusionary.

A moderate or severe exacerbation of COPD ending within 6 weeks prior to dosing (Day 1). The end date of an exacerbation is the last day of treatment with systemic corticosteroids or antibiotics.

Prior pulmonary resection or Lung Volume Reduction Surgery [i.e., lobectomy, bronchoscopic lung volume reduction (endobronchial blockers, airway bypass, endobronchial valves, thermal vapor ablation, biological sealants, and airway implants)].

* Cardiovascular Patients with significant or unstable ischemic heart disease, arrhythmia, cardiomyopathy, heart failure (including significant cor pulmonale), uncontrolled hypertension as defined by the Investigator, or any other relevant cardiovascular disorder as judged by the Investigator.
* Current cancer diagnosis requiring treatment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
The percentage (%) emitted dose of radiolabelled BGF MDI deposited in the lungs following a maximal breath-hold of up to 10 s. | Day 1
  Percentage of BGF MDI deposited in the lungs.

SECONDARY OUTCOMES:
Regional airway deposition ratios including the non-normalized parameters O/I and C/P regions and the normalized parameters PI and sC/P of the radiolabelled BGF MDI following a maximal breath-hold of up to 10 s. | Day 1
  Percentages of BGF MDI deposited in different regions of lungs.

OTHER OUTCOMES:
The fraction of the dose of radiolabelled BGF MDI deposited in the oropharyngeal and stomach regions (expressed as % emitted dose) following a maximal breath-hold of up to 10 s. | Day 1
  Percentages of BGF MDI deposited in oropharyngeal and stomach regions.
The fraction of the dose of radiolabelled BGF MDI deposited on the actuator (expressed as % ex-valve dose) and exhalation filter (expressed as % emitted dose) following a maximal breath-hold of up to 10 s. | Day 1
  Percentages of BGF MDI deposited on the actuator and exhalation filter."
Adverse Events | Up to 14 days
  Number and percentage of patients with at least one treatment emergent adverse events (TEAEs) will be reported. In addition, the number and % of patients reporting TEAEs will be tabulated by maximum intensity and maximum reported causality to investigation product within a patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ezanul Wahab, Principal Investigator — Simbec Research
Locations (2):
- United Kingdom (2):
  - Research Site, Llanelli
  - Research Site, Merthyr Tydfil

REFERENCES:
- [Derived] Usmani O, Roche N, Wahab E, Israel S, Jenkins M, Trivedi R, Dorinsky P, Aurivillius M. A scintigraphy study of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler in patients with moderate-to-very severe chronic obstructive pulmonary disease. Respir Res. 2021 Oct 7;22(1):261. doi: 10.1186/s12931-021-01813-w. PMID 34620167